CLINICAL TRIAL: NCT07161817
Title: Effect of Semirecumbent and Lateral Positioning on Postoperative Hypoxemia : a Randomized Controlled Trial
Brief Title: Effect of Postural Changes on Postoperative Hypoxemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuhu Ma (Other)
Responsible Party: Sponsor-Investigator, Yuhu Ma, Doctor, LanZhou University
Organization: LanZhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Postoperative Hypoxemia
Record Dates: First submitted 2025-08-23; First posted 2025-09-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Hypoxemia; Position Differences
Keywords: Lateral positioning; Hypoxemia; Semirecumbent positioning
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semirecumbent positioning (Experimental): Patients in the Semirecumbent positioning were placed in the bed and the head of the bed was raised by 30 °, allowing flexibility based on patient comfort and surgical requirements.
  Interventions: Behavioral: Semirecumbent positioning
- Lateral positioning (Experimental): Patients allocated to lateral positioning were placed at 90° on a horizontal bed, supported with a pillow to maintain neutral alignment of the spine and avoid hyperextension or forward flexion of the neck. No preference was specified for left or right lateral decubitus positioning, allowing flexibility based on patient comfort and surgical requirements.
  Interventions: Behavioral: Lateral positioning

INTERVENTIONS:
Behavioral: Lateral positioning — Patients allocated to lateral positioning were placed at 90° on a horizontal bed, supported with a pillow to maintain neutral alignment of the spine and avoid hyperextension or forward flexion of the neck. No preference was specified for left or right lateral decubitus positioning, allowing flexibility based on patient comfort and surgical requirements.
  Arms: Lateral positioning
Behavioral: Semirecumbent positioning — Patients in the semi-recumbent position were placed in the bed and the head of the bed was raised by 30 °, allowing flexibility based on patient comfort and surgical requirements.
  Arms: Semirecumbent positioning

SUMMARY:
The goal of this clinical trial is to learn which positioning strategy works better to prevent postoperative hypoxemia in surgical patients: semirecumbent positioning or lateral positioning. It will also learn about the safety and effectiveness of these two positioning approaches. The main questions it aims to answer are:

Does semirecumbent positioning reduce the incidence of postoperative hypoxemia more effectively than lateral positioning? Does lateral positioning reduce the incidence of postoperative hypoxemia more effectively than semirecumbent positioning? What are the differences in patient comfort and recovery outcomes between these two positioning strategies? Researchers will compare semirecumbent positioning directly to lateral positioning to see which approach is more effective in preventing postoperative hypoxemia.

Participants will:

Be randomly assigned to either semirecumbent positioning or lateral positioning after surgery Have their oxygen levels and breathing monitored regularly during the postoperative period Receive standard post-surgical care with their assigned positioning strategy Be assessed for comfort levels and any positioning-related complications Have their recovery progress tracked throughout their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above and 80 or below who received general anesthesia and intubation

Exclusion Criteria:

Inclusion criteria:

- Patients aged 18 years and above, and 80 years and below, who received general anesthesia and intubation;

Exclusion criteria:

* Presence of hypotension or bradycardia upon entering the anesthesia recovery room;
* Preoperative hypoxemia;
* Surgical procedures where body position adjustment is not possible or is prohibited due to the nature of the surgery;
* Surgical procedures involving severe cardiovascular or cerebrovascular diseases, severe pulmonary diseases, intracranial hypertension, etc.;
* Intubation more than 3 times.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxaemia | Within 24 hours after the surgery was completed
  Defined as any occurrence of oxygen saturation (SpO2) ≤90% for at least five seconds during the initial 10 minute period after positioning.

SECONDARY OUTCOMES:
Rrequency of airway rescue interventions | Within 24 hours after the surgery was completed
  Increased oxygen flow, jaw thrust manoeuvre, mask ventilation
incidence of severe hypoxaemia | Within 24 hours after the surgery was completed
  oxyhemoglobin saturation ≤85%
Lowest oxygen saturation | Within 24 hours after the surgery was completed
  Defined as the oxygenation nadir during 10 minutes of continuous measurement.
Duration of stay in the post-anaesthesia care | Perioperative/Periprocedural
  Duration of stay in the post-anaesthesia care
wound pain | Perioperative/Periprocedural
  VAS scale was used to measure pain intensity. The VAS uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. A VAS score between 4-7 represents "mild pain", a score between 4-7 represents "moderate pain" and a score between 8-10 represents "severe pain".
Adverse events | Perioperative/Periprocedural
  hypotension, arrhythmia, and some other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yatao Liu, Doctor, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Guo K, Sun J, Yang Y, Wu Y, Tang X, Xu Y, Chen Q, Zeng S, Wang L, Liu S. Semirecumbent Positioning During Anesthesia Recovery and Postoperative Hypoxemia: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2416797. doi: 10.1001/jamanetworkopen.2024.16797. PMID 38941098
- [Result] Ye H, Chu LH, Xie GH, Hua YJ, Lou Y, Wang QH, Xu ZX, Tang MY, Wang BD, Hu HY, Ying J, Yu T, Wang HY, Wang Y, Ye ZJ, Bao XF, Wang MC, Chen LY, Wang XX, Zhang XB, Huang CS, Wang J, Lu YP, Luo FQ, Zhou W, Wang CG, Cheng H, Liu WJ, Luo J, Wu YQ, Li RR, Wang D, Hou LQ, Shi L, Zhang J, Wang K, Pi X, Zhou R, Yang QQ, Wan PL, Li H, Wu SJ, Song SW, Cui P, Shu L, Islam N, Fang XM. Effect of lateral versus supine positioning on hypoxaemia in sedated adults: multicentre randomised controlled trial. BMJ. 2025 Aug 19;390:e084539. doi: 10.1136/bmj-2025-084539. PMID 40829895